CLINICAL TRIAL: NCT00273468
Title: A Randomised, Active Control, Double-blind, Double-dummy, Parallel-group, Multi-national Study to Assess the Efficacy, Tolerability and Safety of the Granisetron Transdermal Delivery System in Chemotherapy-induced Nausea and Vomiting (CINV) Associated With the Administration of Moderately or Highly Emetogenic Multi-day Chemotherapy
Brief Title: To Study the Safety and Effectiveness of a Granisetron Patch to Treat Chemotherapy-Induced Nausea and Vomiting (CINV)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Kyowa Kirin Co., Ltd. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 392MD/15/C
Record Dates: First submitted 2006-01-06; First posted 2006-01-09 (Estimated); Last update posted 2024-06-17 (Actual); Status verified 2024-06

CONDITIONS: Chemotherapy-induced Nausea and Vomiting
MeSH Terms: conditions — Vomiting | interventions — Granisetron

INTERVENTIONS:
Drug: Granisetron

SUMMARY:
To study the safety and effectiveness of a granisetron patch to treat Chemotherapy-Induced Nausea and Vomiting (CINV)

ELIGIBILITY:
Inclusion Criteria:

* Patients must be of non-childbearing potential and female patients must have a negative pregnancy test at the Screening Visit
* Histologically and/or cytologically confirmed cancer with ECOG ≤2
* Life expectancy of ≥ 3 months
* Assigned to receive the first cycle of a new multi-day chemotherapy regimen including the daily administration of cytotoxic agent(s) with the emetogenic potential of level 3-5 (Hesketh Classification) on 3-5 days

Exclusion Criteria:

* Hypersensitivity to adhesive plasters
* Contraindications to 5-HT3 receptor antagonists
* Clinically relevant abnormal laboratory values or hepatic, renal, infectious, neurological or psychiatric disorders or any other major systemic illness at the discretion of the Investigator
* Any cause for nausea and vomiting other than CINV
* Clinically relevant abnormal ECG parameters
* Concomitant radiotherapy of total body, brain or upper abdomen within one week of study entry or planned during the study
* A patient taking a medication to control the symptoms of a brain tumour, brain metastasis or seizure disorder

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 630
Dates: Start 2006-01; Study Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
Percentage of patients achieving Complete Control of CINV from the first administration until 24 h after the last administration of the moderately or highly emetogenic chemotherapy

SECONDARY OUTCOMES:
Times from start of chemotherapy to treatment failure for complete control (CC) and complete response (CR)
Time from start of chemotherapy to first administration of rescue medication
Time from start of chemotherapy to first emetic episode (vomiting/retching)
Percentage of patients achieving CC and CR of CINV during different time periods
Adverse events collected until 14 days after patch removal
Patch adhesion

REFERENCES:
- [Derived] Boccia RV, Gordan LN, Clark G, Howell JD, Grunberg SM; Sancuso Study Group. Efficacy and tolerability of transdermal granisetron for the control of chemotherapy-induced nausea and vomiting associated with moderately and highly emetogenic multi-day chemotherapy: a randomized, double-blind, phase III study. Support Care Cancer. 2011 Oct;19(10):1609-17. doi: 10.1007/s00520-010-0990-y. Epub 2010 Sep 12. PMID 20835873